CLINICAL TRIAL: NCT07390045
Title: Exercise and Cognitive Rehabilitation Interventions for Older Cancer Survivors: A Pilot Randomized Controlled Trial
Brief Title: Exercise and Cognitive Rehabilitation Interventions for Older Cancer Survivors
Acronym: ECO 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC26001
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: geriatric oncology; cancer survivors; exercise; cognitive rehabilitation; cognition
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise for Cancer Patients (EXCAP; Intervention) (Experimental): Exercise for Cancer Patients (EXCAP) is an individually tailored, low-to-moderate intensity, home-based walking and progressive resistance exercise program designed for patients with cancer delivered by an exercise physiologist. It also includes digital health applications, allowing the tracking of exercise adherence, barriers to exercise, and symptoms.
  Interventions: Behavioral: EXCAP
- Memory and Attention Adaptation Training (MAAT; Intervention) (Experimental): Memory and Attention Adaptation Training (MAAT) is an intervention based on cognitive behavioral therapy principles that integrates cognitive rehabilitation skills and provides education and training in adaptive behavioral coping skills, stress management techniques, and compensation strategies to address CRCD.
  Interventions: Behavioral: MAAT
- Usual Care (No Intervention): Patients in the control group will receive care as usual.
- Exercise and Cognition (ECO; Intervention) (Experimental): Patients will receive the integrated EXCAP and MAAT interventions.
  Interventions: Behavioral: ECO

INTERVENTIONS:
Behavioral: EXCAP — The first component of the EXCAP exercise program is an individually tailored walking prescription and provides low to moderately intense aerobic exercise [5-8 exercise rating of perceived exertion on the American College of Sports Medicine (ACSM) revised rating scale, which is a visual analog scale ranging from 1 = "Not tired at all" to 10 = "So tired, I can't go anymore"] 7 days a week. This walking prescription will be developed and individually tailored for each patient based on step data reported by the patient. A Garmin activity tracker (a wearable sensor-based device) will be used to record the number of steps they walk daily during the 4-7 day baseline assessment. Patients will report their steps daily on a paper form, electronically via REDCap, or over the phone to the study staff at the end of the 4-7 day baseline assessment period. Alternatively, steps can also be obtained via the activity tracker by study staff.
  Arms: Exercise for Cancer Patients (EXCAP; Intervention)
Behavioral: MAAT — The MAAT intervention consists of 10 manualized workshops that will be delivered by a trained clinician. Patients will be provided with a workbook for skills practice in between sessions. A summary of workshop content is provided in Table 1.
  During Workshop #2, study staff or a trained clinician will provide patients with a link to a Vimeo video through the app. The Vimeo video has been created by the study team and guides patients through relaxation strategies to use before stressful events. Patients will be able to access the video without providing any personal information to the website.
  Arms: Memory and Attention Adaptation Training (MAAT; Intervention)
Behavioral: ECO — Patients will receive the integrated EXCAP and MAAT interventions.
  Arms: Exercise and Cognition (ECO; Intervention)

SUMMARY:
The objective of this study is to assess the preliminary effects of an integrated exercise and cognitive rehabilitation intervention (ECO), an exercise intervention (EXCAP), and a cognitive rehabilitation intervention (MAAT) as compared to usual care on objective cognition (Trail Making Test).

DETAILED DESCRIPTION:
Cancer-Related Cognitive Dysfunction (CRCD) is a prevalent problem for older cancer survivors. Sixty-four percent of current cancer survivors are aged ≥65, and by 2040, it is estimated that over 19 million older cancer survivors will be living in the United States. Up to 50% of these individuals experience CRCD post-treatment, which can persist for years after treatment completion. For older adults, CRCD can affect their ability to perform daily tasks, such as taking medications or managing finances, reducing their overall independence. Although evidence-based interventions exist to treat CRCD, older adults were underrepresented in these trials, despite them being most at risk for CRCD and its consequences. The National Cancer Institute, topic experts, and patient advocates have highlighted the urgent need for accessible interventions to address CRCD symptoms, particularly for older adults.

Exercise for Cancer Patients (EXCAP) is an individually tailored, low-to-moderate intensity, home-based walking and progressive resistance exercise program designed for patients with cancer delivered by an exercise physiologist. The Investigators adapted EXCAP for digital health applications, allowing the tracking of exercise adherence, barriers to exercise, and symptoms. In a large randomized controlled trial (RCT), EXCAP improved patient-reported cognition compared to usual care. In older adults with cancer, EXCAP patients demonstrated improvements in cognitive impairment, as assessed via the Trail-Making Test, which evaluates processing speed.

Memory and Attention Adaptation Training (MAAT) was previously shown to improve CRCD and psychological function in three clinical trials. The Investigators tailored aspects for the particular needs of older adults, including support for telehealth delivery. The intervention, based on cognitive behavioral therapy principles, integrates cognitive rehabilitation skills and provides education and training in adaptive behavioral coping skills, stress management techniques, and compensation strategies to address CRCD. MAAT is standardized via a manual and delivered one-on-one via video-conferencing over 10 weekly workshops by a trained clinician. In a pilot RCT, MAAT improved perceived cognition [Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) and objective cognition (e.g., processing speed). In a separate study of 34 older adults with cancer, improvements from baseline to post-intervention were observed in objective cognitive measures and perceived cognition.

Exercise and Cognition (ECO) leverages the synergy between EXCAP and MAAT, and enhances both general and exercise self-efficacy, improves adherence, and promotes lasting behavior change for sustained cognitive benefits. Adapted with input from the patient advisory board, ECO is a 12-week program delivered virtually by an exercise physiologist and a trained clinician, facilitated through digital health applications. Delivering both interventions simultaneously was evaluated in a single-arm pilot study of eight older adults with cancer who had completed curative treatments and were experiencing residual CRCD symptoms. Preliminary results suggest greater self-efficacy and exercise adherence. From baseline to post-intervention, all patients reported clinically meaningful improvements in FACT-Cog; these improvements were greater than those observed with EXCAP or MAAT intervention alone.

However, it is unknown which behavioral intervention is most effective at addressing CRCD symptoms. It is also unknown which type of CRCD intervention is the "best fit" for each patient. To inform the design of a future R01-funded definitive RCT to fill these gaps, the Investigators need to obtain more precise estimates of ECO's effects and identify the most appropriate comparison arms.

ELIGIBILITY:
Inclusion criteria:

* Age ≥65 years (from date of consent, confirmed on the electronic medical record)
* A diagnosis of any cancer
* Have completed curative intent treatments

  * Patients on endocrine therapies are allowed to enroll
  * Patients with hematologic malignancies after autologous or allogeneic stem cell transplant are allowed to enroll if they have completed curative-intent treatment
* Answered "yes" to the verbal question "Do you have concerns about memory or other thinking abilities following your cancer treatment?"
* Able to speak English (interventions are available in English only)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3#
* No medical contraindications to exercise#
* Able to walk 4 meters#
* Able to provide informed consent#

  * Confirmed through eligibility confirmation with the patient's oncologist or their designee

Exclusion criteria:

* Any physical, psychological, or social impairments that would interfere with a patient's ability to participate in the study as determined by the patient's oncologist or their designee
* Unwilling to complete study procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective cognition | Change from baseline to week 12
  Trail Making Test A & B: The Trail Making Test assesses sustained attention. The Written Trail Making Test A & B is preferred; however, if this is not feasible, the oral Trail Making Test will be utilized. There is not a range, lower scores indicating better performance

SECONDARY OUTCOMES:
Perceived Cognition | Change from baseline to week 12
  Functional Assessment of Cancer Therapy-Cognition Perceived Cognitive Abilities. Scores range from 0-28, higher scores are better.
Depressive symptoms | Change from baseline to week 12
  Center for Epidemiological Studies Depression Scale (CES-D): The CES-D is a 20-item depression scale developed and validated for use with various populations. Scores range from 0-60, higher scores are worst.
Anxiety symptoms | Change from baseline to week 12
  General Anxiety Disorder-7 (GAD-7): GAD-7 is a 7-item screening tool for anxiety. Scores range from 0-21, higher scores are worst.

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators if requested. Published papers will be made available in portable document format.
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years after study completion

REFERENCES:
- [Background] Loh KP, Sanapala C, Watson EE, Jensen-Battaglia M, Janelsins MC, Klepin HD, Schnall R, Culakova E, Vertino P, Susiarjo M, Lin PJ, Mendler JH, Liesveld JL, Huselton EJ, Taberner K, Mohile SG, Mustian K. A single-arm pilot study of a mobile health exercise intervention (GO-EXCAP) in older patients with myeloid neoplasms. Blood Adv. 2022 Jul 12;6(13):3850-3860. doi: 10.1182/bloodadvances.2022007056. PMID 35320340
- [Background] Loh KP, Sanapala C, Janelsins M, Klepin HD, Schnall R, Culakova E, Sohn MB, Vertino P, Susiarjo M, Jensen-Battaglia M, Becker MW, Liesveld J, Mendler JH, Huselton E, Lin PJ, Mustian K. Protocol for a pilot randomized controlled trial of a mobile health exercise intervention for older patients with myeloid neoplasms (GO-EXCAP 2). J Geriatr Oncol. 2022 May;13(4):545-553. doi: 10.1016/j.jgo.2021.12.011. Epub 2021 Dec 21. PMID 34949540